CLINICAL TRIAL: NCT02754596
Title: Prospective, Randomized Phase II Study Comparing Two Elution Rates of Glaukos Travoprost Intraocular Implants to Timolol Maleate Ophthalmic Solution, USP 0.5%
Brief Title: Study Comparing Travoprost Intraocular Implants to Timolol Ophthalmic Solution
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GC-009
Record Dates: First submitted 2016-03-15; First posted 2016-04-28 (Estimated); Results first posted 2023-08-09 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Glaucoma Open-angle
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Travoprost Intraocular Implant, high elution (Experimental): This implant will be surgically implanted and elute travoprost, a prostaglandin.
  Interventions: Drug: Travoprost Intraocular Implant, high elution
- Travoprost Intraocular Implant, low elution (Experimental): This implant will be surgically implanted and elute travoprost, a prostaglandin.
  Interventions: Drug: Travoprost Intraocular Implant, low elution
- Timolol Maleate Ophthalmic Solution, 0.5% (Active Comparator): Timolol, a beta blocker, will be dosed twice daily
  Interventions: Drug: Timolol Maleate Ophthalmic Solution, 0.5%

INTERVENTIONS:
Drug: Travoprost Intraocular Implant, high elution — Surgical implant placed within the eye to elute travoprost.
  Arms: Travoprost Intraocular Implant, high elution
Drug: Travoprost Intraocular Implant, low elution — Surgical implant placed within the eye to elute travoprost
  Arms: Travoprost Intraocular Implant, low elution
Drug: Timolol Maleate Ophthalmic Solution, 0.5% — Instillation of one drop of timolol in the study eye twice daily
  Arms: Timolol Maleate Ophthalmic Solution, 0.5%

SUMMARY:
This is a randomized trial comparing two elution doses of the Travoprost Intraocular implant to timolol ophthalmic solution.

DETAILED DESCRIPTION:
This is a randomized trial comparing two elution doses of the Travoprost Intraocular implant to timolol ophthalmic solution in patients with open-angle glaucoma. Study assessments will include IOP and medication use as well as safety parameters.

ELIGIBILITY:
Inclusion Criteria:

* Open angle glaucoma

Exclusion Criteria:

* Uveitic, neovascular, or angle closure glaucoma; or glaucoma associated with vascular disorders.
* Functionally significant visual field loss, including severe nerve fiber bundle defects.
* Prior glaucoma surgery.
* Uncontrolled systemic disease, pregnant females or those planning a pregnancy.
* Other ocular status conditions, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2016-03-29 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2020-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Stephens, O.D., Study Chair — Glaukos Corporation
Locations (1):
- John Berdahl, MD, Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No
The datasets generated during and/or analyzed during the current study are not publicly available at this time due to ongoing U.S. Food and Drug Administration review of a New Drug Application for the travoprost intraocular implant.

REFERENCES:
- [Derived] Berdahl JP, Sarkisian SR Jr, Ang RE, Doan LV, Kothe AC, Usner DW, Katz LJ, Navratil T; Travoprost Intraocular Implant Study Group. Efficacy and Safety of the Travoprost Intraocular Implant in Reducing Topical IOP-Lowering Medication Burden in Patients with Open-Angle Glaucoma or Ocular Hypertension. Drugs. 2024 Jan;84(1):83-97. doi: 10.1007/s40265-023-01973-7. Epub 2023 Dec 7. PMID 38060092

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects underwent a washout from IOP-lowering medications after enrollment and prior to assignment to groups
Period: Overall Study
Arm/Group | Travoprost Intraocular Implant, High Elution | Travoprost Intraocular Implant, Low Elution | Timolol Maleate Ophthalmic Solution, 0.5%
Started | 51 | 54 | 49
Month 3 | 51 | 54 | 49
Completed | 44 | 46 | 45
Not Completed | 7 | 8 | 4
Not completed — Withdrawal by Subject | 3 | 4 | 0
Not completed — Physician Decision | 1 | 1 | 1
Not completed — Lost to Follow-up | 1 | 1 | 2
Not completed — Death | 0 | 2 | 0
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Other | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Each participant received treatment in only one eye
Groups:
- Total: Total of all reporting groups
Arm/Group | Travoprost Intraocular Implant, High Elution | Travoprost Intraocular Implant, Low Elution | Timolol Maleate Ophthalmic Solution, 0.5% | Total
Number analyzed (Participants) | 51 | 54 | 49 | 154
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 30 | 24 | 82
  >=65 years | 23 | 24 | 25 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (9.8) | 61.4 (13.9) | 63.0 (12.6) | 62.7 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 29 | 20 | 76
  Male | 24 | 25 | 29 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 3 | 8
  Not Hispanic or Latino | 47 | 53 | 46 | 146
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 5 | 6 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 8 | 5 | 19
  White | 41 | 41 | 37 | 119
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Baseline IOP [Mean (Standard Deviation); unit: mmHg] — Baseline IOP in mmHg was measured at 8AM by Goldmann tonometry after the appropriate washout from IOP-lowering medication(s) used at Screening
  mmHg | 26.4 (4.9) | 25.3 (4.7) | 25.3 (3.9) | 25.7 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: IOP (mmHg) Change From Baseline at Week 12
Description: Change from baseline in IOP (measured in mmHg) at week 12. Negative values represent reductions in IOP from baseline.
Time Frame: 12 weeks
Population: intent-to-treat population
Measure: Mean (Standard Error); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Travoprost Intraocular Implant, High Elution | Travoprost Intraocular Implant, Low Elution | Timolol Maleate Ophthalmic Solution, 0.5%
Number analyzed (Participants) | 51 | 54 | 49
Number analyzed (eyes) | 51 | 54 | 49
mmHg | -8.3 (0.34) | -7.7 (0.26) | -7.5 (0.21)

2. Other Pre Specified Outcome: Severe Adverse Events
Description: The number and percent of subjects with severe adverse events in the study eye
Time Frame: Post-op through Month 36
Population: study eyes
Measure: Count of Participants; unit: Participants
Arm/Group | Travoprost Intraocular Implant, High Elution | Travoprost Intraocular Implant, Low Elution | Timolol Maleate Ophthalmic Solution, 0.5%
Number analyzed (Participants) | 51 | 54 | 49
Participants | 2 | 2 | 2

ADVERSE EVENTS:
Time Frame: overall study period of 36 months
Arm/Group | Travoprost Intraocular Implant, High Elution | Travoprost Intraocular Implant, Low Elution | Timolol Maleate Ophthalmic Solution, 0.5%
All-Cause Mortality (participants affected / at risk) | 0/51 | 2/54 | 0/49
Serious Adverse Events (participants affected / at risk) | 4/51 | 9/54 | 3/49
Other Adverse Events (participants affected / at risk) | 28/51 | 22/54 | 14/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Travoprost Intraocular Implant, High Elution (N=51) | Travoprost Intraocular Implant, Low Elution (N=54) | Timolol Maleate Ophthalmic Solution, 0.5% (N=49)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
cardiac disorders (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
death (General disorders) | 0 (0) | 2 (2) | 0 (0)
pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
myasthenia gravis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Travoprost Intraocular Implant, High Elution (N=51) | Travoprost Intraocular Implant, Low Elution (N=54) | Timolol Maleate Ophthalmic Solution, 0.5% (N=49)
cataract (Eye disorders) | 4 (4) | 3 (3) | 1 (1)
visual acuity reduced (Eye disorders) | 3 (3) | 4 (4) | 1 (1)
vitreous detachment (Eye disorders) | 2 (2) | 3 (3) | 1 (1)
blepharitis (Eye disorders) | 3 (3) | 1 (1) | 1 (1)
conjunctival hemorrhage (Eye disorders) | 2 (2) | 3 (3) | 0 (0)
eye pain (Eye disorders) | 3 (3) | 0 (0) | 1 (1)
foreign body sensation in eyes (Eye disorders) | 1 (1) | 3 (3) | 0 (0)
eye inflammation (Eye disorders) | 3 (3) | 0 (0) | 0 (0)
bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 3 (3)
arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 0 (0)
intraocular pressure increased (Investigations) | 2 (2) | 2 (2) | 5 (5)
hypertension (Vascular disorders) | 2 (2) | 4 (4) | 1 (1)
drug hypersensitivity (Immune system disorders) | 2 (2) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of data from this study.

DOCUMENTS (2):
  • Study Protocol (2016-09-16): https://cdn.clinicaltrials.gov/large-docs/96/NCT02754596/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-06): https://cdn.clinicaltrials.gov/large-docs/96/NCT02754596/SAP_001.pdf